CLINICAL TRIAL: NCT02505100
Title: Impact of Complementary Medicine Techniques (Therapeutic Touch and Hypno Analgesia) on the Term of Delivery of Patients Hospitalized for Preterm Labor (Hypnorelax)
Acronym: Hypnorelax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHRIP 1439287N
Record Dates: First submitted 2015-07-02; First posted 2015-07-22 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2018-02

CONDITIONS: Premature Birth
Keywords: threat of premature birth
MeSH Terms: conditions — Premature Birth | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Touching relaxant (Experimental): session of massage
  Interventions: Other: Touching relaxant
- Hypnoses (Experimental): session of hypnoses
  Interventions: Other: Hypnoses
- Standared care (No Intervention): standard care

INTERVENTIONS:
Other: Touching relaxant
  Arms: Touching relaxant
Other: Hypnoses
  Arms: Hypnoses

SUMMARY:
The threat of premature birth (MAP) is the leading cause of hospitalization during pregnancy complicated by preterm delivery in 5-10% of cases in developed countries. Psychological stress that encompasses anxiety and anxiety resounding including sleep quality can be a work of preacher and premature delivery.

Preterm birth before 37 has an impact on the survival and health of the newborn. It is the leading cause of mortality and obstetric complications. It has a cost both for the newborn, the term parturient health but also the financial cost by the management before delivery and the consequences of a premature birth.

The usual management of MAP is hospitalized with tocolysis, monitoring and rest. The hospitalization and invasive procedures contribute to increasing stress. It therefore seems necessary to seek to diversify and master reputable techniques for their effectiveness on mastering stress and improving sleep quality as hypnosis and feel relaxing.

Hypnosis in obstetrics is used primarily to control pain, nausea and postpartum depression. It also reduces preoperative anxiety and during induction of anesthesia, as well as behavioral disorders during the first postoperative week. Hypnosis can play an important role in the prevention of preterm birth. In a non-randomized study, hypnosis combined with drug therapy has prolonged pregnancy of patients followed in high risk pregnancy.

The relaxing touch brings relaxation and well being. In obstetrics, it has an influence on the anti-stress hormones and plays a role in reducing pain during childbirth.

Few studies interested in hypnosis and relaxation therapies in pregnant women, especially in case of MAP. The published data relate to a small number of patients and a low level of evidence. Although there seems promising results, prospective studies are needed to conclude its effectiveness in improving the stress, pain or other parameters.

Health workers trained in these techniques could observe during their production improved sleep disorders, stress, better communication between doctor and patient. Moreover, these treatments could induce an improvement in the overall care of patients, and therefore have an impact on the continuation of pregnancy.

These findings are based on these hypothesis. There is a clinical gain the contribution of hypnosis and relaxing touch in women hospitalized for MAP before 32 weeks of gestation. This would, among other improvements in sleep disorders and stress, decrease pain, and acting on the extension of the term of pregnancy in women followed by these techniques and a decrease in hospitalizations of newborns premature neonatology and neonatal intensive care units.

DETAILED DESCRIPTION:
The threat of premature birth (MAP) is the leading cause of hospitalization during pregnancy complicated by preterm delivery in 5-10% of cases in developed countries. Psychological stress that encompasses anxiety and anxiety resounding including sleep quality can be a work of preacher and premature delivery.

Preterm birth before 37 has an impact on the survival and health of the newborn. It is the leading cause of mortality and obstetric complications. It has a cost both for the newborn, the term parturient health but also the financial cost by the management before delivery and the consequences of a premature birth.

The usual management of MAP is hospitalized with tocolysis, monitoring and rest. The hospitalization and invasive procedures contribute to increasing stress. It therefore seems necessary to seek to diversify and master reputable techniques for their effectiveness on mastering stress and improving sleep quality as hypnosis and feel relaxing.

Hypnosis in obstetrics is used primarily to control pain, nausea and postpartum depression. It also reduces preoperative anxiety and during induction of anesthesia, as well as behavioral disorders during the first postoperative week. Hypnosis can play an important role in the prevention of preterm birth. In a non-randomized study, hypnosis combined with drug therapy has prolonged pregnancy of patients followed in high risk pregnancy.

The relaxing touch brings relaxation and well being. In obstetrics, it has an influence on the anti-stress hormones and plays a role in reducing pain during childbirth.

Few studies interested in hypnosis and relaxation therapies in pregnant women, especially in case of MAP. The published data relate to a small number of patients and a low level of evidence. Although there seems promising results, prospective studies are needed to conclude its effectiveness in improving the stress, pain or other parameters.

Health workers trained in these techniques could observe during their production improved sleep disorders, stress, better communication between doctor and patient. Moreover, these treatments could induce an improvement in the overall care of patients, and therefore have an impact on the continuation of pregnancy.

These findings are based on these hypothesis. There is a clinical gain the contribution of hypnosis and relaxing touch in women hospitalized for MAP before 32 weeks of gestation. This would, among other improvements in sleep disorders and stress, decrease pain, and acting on the extension of the term of pregnancy in women followed by these techniques and a decrease in hospitalizations of newborns premature neonatology and neonatal intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Patient hospitalized for the first time for MAP (preterm labor) at the Robert Debré hospital as defined in CNGOF (National college of French gynecologists and obstetricians):

  * frequent and regular uterine contractions (at least 3 in 30 minutes)
  * significant cervical changes,
  * before 37 weeks of amenorrhea (SA).
* Single or multiple pregnancies
* Age greater than or equal to 18 years
* Patient between 24 + 0 and 32 + 0 weeks of gestation.
* Patient not opposing its participation
* Patient beneficiary of a social security

Exclusion Criteria:

* Not understanding of technology (language barrier ...)
* Psychiatric Pathology (cons-indication to hypnosis: schizophrenia, paranoia)
* Refusal by the patient
* Age <18 years

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of weeks of gestation | 4 months
  Term of delivery will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Céline Perrudin, Principal Investigator — APHP
Locations (1):
- Perrudin, Paris, France